CLINICAL TRIAL: NCT07135583
Title: Non-Invasive Interventions and Biomarker Identification for Respiratory Recovery in Chronic Spinal Cord Injury
Brief Title: Non-Invasive Interventions for Respiratory Recovery in Chronic Spinal Cord Injury
Acronym: Combinatorial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Jayakrishnan Nair, Assistant Professor, Thomas Jefferson University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRBID-2023-1796; 1349389 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injury, Chronic; Spinal Cord Injury Cervical; Spinal Cord Injury Thoracic; Incomplete Spinal Cord Injury
Keywords: "Spinal Cord Stimulation" [MeSH]; acute intermittant hypoxia; respiratory resistance training; Genetic Biomarker; Blood biomarker
MeSH Terms: conditions — Spinal Cord Injuries; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: A Single-blind, placebo-controlled, randomized order, William Latin cross-over experimental design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combined Intervention (Experimental): Experimental Combination of HiCO2-AIH+ tSCS paired respiratory exercise
  Interventions: Other: Active Comparator: Single Intervention 1; Other: Active Comparator: Single Intervention 2; Behavioral: Respiratory Resistance Exercise
- Single Intervention 1 (Active Comparator): Combination of HiCO2-AIH+ Sham stimulation paired respiratory exercise
  Interventions: Other: Active Comparator: Single Intervention 1; Behavioral: Respiratory Resistance Exercise
- Single Intervention 2 (Active Comparator): Combination of Sham Exposure + tSCS paired respiratory exercise
  Interventions: Other: Active Comparator: Single Intervention 2; Behavioral: Respiratory Resistance Exercise
- Sham Intervention (Placebo Comparator): Combination of Sham Exposure + Sham Stimulation paired respiratory exercise
  Interventions: Behavioral: Respiratory Resistance Exercise

INTERVENTIONS:
Other: Active Comparator: Single Intervention 1 — Acute intermittent hypercapnic-hypoxia (15 episodes of 1.5 minute O2= 9%, CO2=4% and balance N2, interspaced with 1.5 min room air
  Arms: Combined Intervention; Single Intervention 1
Other: Active Comparator: Single Intervention 2 — An open-loop continuous tSCS stimulation [30 min duration, low frequency (30 Hz), tolerable intensity (~10-15 mA), 400 µsec pulse width, biphasic symmetric waveform] will be delivered using 2 channels: Channel 1- C4-C5 spine; Channel 2- T4 spine; returning electrodes at ASIS.
  Arms: Combined Intervention; Single Intervention 2
Behavioral: Respiratory Resistance Exercise — Respiratory strength training will be conducted using a standard, spring-loaded threshold device while the participant is receiving either tSCS or Sham tSCS. Participants will complete one warm-up set at a pressure threshold approximately 40% of their pre-test outcomes (obtained on day 1 of the corresponding intervention block) for maximal inspiratory and expiratory pressure generation. Following the warm-up, participants will train at a pressure threshold approximately 70% of their pre-test outcomes and will complete three sets of 6-12 repetitions for both inspiratory and expiratory strength training. A training breath will consist of a ~1-2-second sustained effort through the device, separated by 5-10 seconds of quiet breathing. The order of the three sets each of inspiratory or expiratory training will alternate for each of the five daily sessions; the order on day 1 of training will be randomly determined.
  Other Names: Respiratory Strength Training; Inspiratory resistance training; Expiratory resistance training

SUMMARY:
Spinal cord injuries (SCI) can seriously affect a person's ability to breathe. This happens because the injury can damage the nerves that control the muscles used for breathing. As a result, people with SCI often face breathing problems, a higher risk of lung infections, and even early death. While breathing exercises can help strengthen these muscles, they often aren't intense enough to make a big difference, especially in people with long-term injuries.

This research project is exploring a new way to improve breathing in people with chronic SCI. The goal is to "wake up" the remaining nerve pathways that still connect the brain and spinal cord to the breathing muscles. By doing this, the investigators hope to make breathing exercises more effective and improve overall respiratory health.

The investigators are testing a combination of two non-invasive (non-surgical) techniques:

Transcutaneous Spinal Cord Stimulation (tSCS): This uses small electrical pulses delivered through the skin to stimulate the spinal cord and help activate the muscles used for breathing.

Hypercapnic-Hypoxia Protocol (HiCO₂-AIH): This involves breathing air with lower oxygen and higher carbon dioxide for short periods. This naturally increases the brain's drive to breathe and may help strengthen the breathing muscles.

The investigators believe that using these two techniques together will "prime" the nervous system, making it more responsive to breathing exercises. This could lead to better outcomes for people with SCI.

In addition to testing this treatment, the investigators are also collecting saliva and blood samples to look for biomarkers-biological clues that might help predict who will benefit most from this therapy. These include genetic markers and signs of nerve damage in the blood.

Who Can Participate

The investigators are looking for adults aged 18 to 70 who:

Have had a spinal cord injury for at least one year. Have an injury between the neck and upper back (from C3 to T8). Have an incomplete injury (some nerve function remains). Are medically stable and cleared by a doctor. Have at least a 20% reduction in breathing strength. What Participants Will Do

Each participant will complete four rounds of treatment. Each round includes four days in a row of therapy, followed by a three-week break before the next round.

Each daily session lasts about two hours and includes:

Breathing special air mixtures (low oxygen and high carbon dioxide) for short periods, followed by normal air.

A short break. Then, spinal cord stimulation combined with breathing exercises that use resistance (like breathing through a straw).

What the Investigators Will Measure

The investigators will track:

Breathing ability using lung function tests and pressure measurements. Nerve activity using brain and spinal cord stimulation to see how well the diaphragm (the main breathing muscle) responds.

Safety by monitoring oxygen levels, heart rate, blood pressure, and breathing responses during each session.

Biological Samples

Participants will provide:

A one-time saliva sample for genetic testing. A one-time blood sample to look for markers of nerve injury. Why This Matters

This study could lead to new, non-invasive treatments that improve breathing and quality of life for people living with spinal cord injuries. By identifying who is most likely to benefit from this therapy, the investigators can also move toward more personalized and effective care in the future.

DETAILED DESCRIPTION:
The overall objectives of this study are:

To determine whether combining hypercapnic-hypoxia protocol (HiCO₂-AIH) and transcutaneous spinal cord stimulation (tSCS) can enhance the effects of respiratory resistance training in individuals with chronic spinal cord injury (SCI).

To explore whether genetic and blood-based biomarkers can help predict how individuals respond to this combined intervention.

We will test these objectives in adults with chronic SCI using a Williams cross-over design. The study will include 16 participants (with statistical power >0.8 and α=0.05), accounting for a 20% dropout rate, for a total enrollment of 20 participants.

Specific Aims

Aim 1:

To determine whether four consecutive days of combined HiCO₂-AIH and tSCS will improve the effectiveness of respiratory resistance training compared to either intervention alone.

Outcomes (measured from PRE to 1 day POST intervention):

Primary Outcome: Change in mouth occlusion pressure at 0.1 seconds (P0.1). Secondary Outcomes: Maximal inspiratory and expiratory pressure generation, forced vital capacity (FVC), neurophysiological measures of cortico-spinal drive (amplitude of transcranial magnetic stimulation [TMS]) and local spinal excitability (amplitude of cervical magnetic stimulation [CMS]) in the diaphragm.

Safety Outcomes: Continuous monitoring of respiratory parameters (end tidal oxygen [O₂] and carbon dioxide [CO₂] concentration, oxygen saturation [SpO₂]) and cardiovascular parameters (blood pressure [BP], heart rate [HR], and electrocardiogram [ECG]) during each session.

Aim 2:

To identify predictive factors for treatment response to the combined HiCO₂-AIH and tSCS intervention using:

1. Genetic polymorphisms related to intermittent hypoxia signaling pathways.
2. Molecular markers of neurotrauma and inflammation found in blood extracellular vesicles (EVs).

Outcomes:

Regression analyses will be conducted to examine the relationship between treatment outcomes and:

Specific genetic single nucleotide polymorphisms (SNPs). Blood-based molecular markers of neurotrauma and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. adults 18 to 70 years of age (the latter to reduce likelihood of cardiovascular disease);
2. chronic SCI for ≥ 1 year at or below C-3 to T-8
3. incomplete SCI based on classification of incomplete-B, C or D
4. medically stable with clearance from physician
5. SCI due to non-progressive etiology
6. >20% impairment in maximal inspiratory or expiratory pressure generation

Exclusion Criteria:

* Individuals will be excluded due to (1) current diagnosis of an additional neurologic condition (eg. multiple sclerosis or stroke) (2) loss of diaphragm EMG activity on forced respiratory tests; (3) severe illness or infection (4) non-healing decubitus ulcers (5) untreated bladder or urinary infections (6) cardiovascular disease (7) lung disease (8) active heterotopic ossification (9) uncontrolled hypertension; (10) severe neuropathic pain; (11) pregnancy (5) severe recurrent and uncontrolled autonomic dysreflexia (6) history of seizure disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
change in mouth occlusion pressure at 0.1 secs (P0.1) | Pre- Baseline (Day 1), Post 1(30 minute post day 4 intervention) and Post 2 ( 24 hours post day 4 intervention)
  It measures the pressure generated at the mouth in the first 0.1 second of inspiration when the airway is unexpectedly occluded at the end of expiration. The negative pressure generation in 0.1 seconds reflects respiratory motor drive without time for modification by sensory systems such as lung stretch or visual input. The inspiratory valve will be occluded prior to the onset of inspiration, without participant awareness, and maintained until the subsequent inspiratory effort. Negative pressure generation will be recorded using a pressure transducer connected to a non-rebreathable mask. All respiratory assessments will be performed in accordance with standard testing guidelines. Measurement indices of ventilation will be obtained using a mouthpiece attached to the pneumotach and nasal clips. The mouth pressure from the pneumotach will be converted to a digital signal using Powerlab C.

SECONDARY OUTCOMES:
Maximum Inspiratory (MIP) & Expiratory (MEP) Pressure | Pre- Baseline (Day 1), Post 1(30 minute post day 4 intervention) and Post 2 ( 24 hours post day 4 intervention)
  Inspiratory pressure generation is indicative of inspiratory strength and is associated with pulmonary health and infection risk. Expiratory pressure generation reflects expiratory respiratory strength and is associated with airway clearance and cough. Inspiratory and expiratory pressure generation improve following weeks of respiratory strength training and after single-day sessions of AIH. Measurements will be obtained using a mouthpiece attached to the pneumotach to measure indices of ventilation, along with the use of nasal clips. To obtain MIP, participants will exhale to residual volume and attempt a maximal inspiration for at least 2 seconds with the inspired line occluded. MEP will be measured with forced expiration against an occluded expired line after the participant inhales to near total lung capacity.
Sniff nasal inspiratory pressure (SNIP) | Pre- Baseline (Day 1), Post 1(30 minute post day 4 intervention) and Post 2 ( 24 hours post day 4 intervention)
  Sniff nasal inspiratory pressure (SNIP) is the measurement of esophageal pressure during maximal sniffs and can be useful in assessing inspiratory muscle strength. To obtain SNIP, the pressure measurement will be obtained through an occluded nostril using a nasal probe, as the participant performs a sniff through the contralateral nostril.
Transcranial Magnetic Stimulation (TMS) evoked Diaphragm Motor Evoked Potentials | Pre- Baseline (Day 1), Post 1(30 minute post day 4 intervention) and Post 2 ( 24 hours post day 4 intervention)
  Subjects will be seated comfortably, fully supported, with their neck slightly flexed. Transcranial magnetic stimulation is performed using a standard technique. The vertex of the skull is identified by the intersection between nasion to inion and tragus to tragus. The region of the cortex responsible for diaphragm motor activation is located approximately 3 cm lateral and 2 cm anterior to the vertex. Single-pulse stimuli are delivered using a handheld double cone coil powered by a magnetic stimulator. The coil is held over the left hemisphere of the brain with current flowing in the anteroposterior direction. The coil is then moved slightly from the pre-determined site and rotated in 45° increments until the largest motor evoked potential (MEP) is observed. This location is marked on a tight-fitting TMS cap placed over the subject's head to ensure accurate coil positioning in future stimulations.
Cervical Magnetic Stimulation (CMS) Diaphragm motor evoked potentials | Pre- Baseline (Day 1), Post 1(30 minute post day 4 intervention) and Post 2 ( 24 hours post day 4 intervention)
  Single-pulse stimuli will be delivered using a handheld circular coil placed over the cervical spine (C7). Recruitment curves are plotted by gradually increasing the intensity of stimulus from 40% to 100% of the maximal stimulator output in 5% increments. Approximately 15 stimulations will be performed at each intensity, separated by 30 seconds. If the subject wishes to take an extended break between stimulations, they may do so until ready to continue.
  As with all procedures, participants will be closely monitored for any discomfort. During these stimulation procedures, subjects will be closely monitored for discomfort and are encouraged to inform the experimenter if they wish to pause testing, take a break, or discontinue stimulations.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Nair, PT, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Center City Campus, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All digital research material included but not limited to images, spreadsheets, protocols, and analysis scripts will be archived and made available via Open Data Commons for Spinal Cord Injury (ODC-SCI) or similar site.
Supporting Information: Study Protocol
Time Frame: The data will be made available within 1 year of the completion of the study (Aug 2028).
Access Criteria: Data on Open Data Commons for Spinal Cord Injury (ODC-SCI) or similar site will be open to public and any researcher